CLINICAL TRIAL: NCT05601739
Title: Interleukin-1β (rs 1143627 T/C) Gene Polymorphism May Increase the Risk of Developing Lumbar Degenerative Disc Disease in Turkish Population: A Preliminary Study
Brief Title: Interleukin-1β (rs 1143627 T/C) Gene Polymorphism May Increase the Risk of Developing LDD in Turkish Population
Status: Completed | Type: Observational
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: YeditepeU-DilekÜ-001
Record Dates: First submitted 2022-07-31; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-07

CONDITIONS: Lumbar Disc Degeneration; Low Back Pain; Inflammation
Keywords: lumbar disc degeneration; polymorphism; interleukin 1 beta; low back pain
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Interleukin 1-β (rs 1143627 T/C) Gene Polymorphism
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lumbar degenerative disc disease: The case group was made of 50 patients, 24 women (48%) and 26 men (52%) with several clinical symptoms suggestive of LDD and the condition confirmed by MRI.
- Healthy: The control group was made of 44 healthy volunteers.

SUMMARY:
This study aims to show the association between the Interleukin-1β (rs 1143627 T/C) gene polymorphism and the patient's pain level, radiological features, functional disability, and spinal flexibility.

DETAILED DESCRIPTION:
Background: Lumbar disc degeneration (LDD), a complex process characterized by phenotypic and genotypic changes, causes low back pain.

Aims: This study aims to show the association between the Interleukin-1β (rs 1143627 T/C) gene polymorphism and the patient's pain level, radiological features, functional disability, and spinal flexibility.

Method: A hospital-based case-control study included 50 LDD patients and 44 healthy controls. In this study, Taqman allelic discrimination analysis was performed for the genotype of the Interleukin-1β (rs 1143627 T/C) gene polymorphism. Differences in Interleukin-1β allele frequencies and genotypes were evaluated between patients and controls. Relationships between allele presence/genotype and disease risk are reported as odds ratios (ORs) with 95% confidence intervals (CIs). The Pfirrmann classification was used to grade the level of disc degeneration on MRI scans, and the McNab's classification was used to classify disc displacements. The pain levels of the patient group were evaluated with VAS and their functional disability with ODI. Spinal flexibility was evaluated using the Modified Schober method and a digital inclinometer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low back pain (over 3 months
* Aged 18-60 years old
* With magnetic resonance imaging (MRI) evidencing LDD with Pfirrmann classification

Exclusion Criteria:

* Cauda equina syndrome
* Lumbar spinal stenosis
* Spinal deformities (scoliosis, kyphosis, spondylolisthesis)
* Vertebral fractures
* Inflammatory rheumatic diseases
* Diabetic neuropathy
* Pregnancy
* Drug and alcohol dependence
* Psychiatric illness
* Oncologic diseases
* Who refuse to sign the consent form and donate a blood sample for analysis of genomic DNA.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study was conducted between April and November 2019. This is a two-centre study undertaken at Yeditepe University Hospital's Department of Neurosurgery and the Yeditepe Institute of Health Sciences Department of Molecular Medicine. One of the analytical research approaches used was a case/control study.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Genotyping - Interleukin-1β (rs 1143627 T/C) gene polymorphism | baseline
  Genotype analysis of interleukin-1β variation was analyzed with Real-Time PCR (polymerase chain reaction) using Applied bioscience 7500 Fast-Real Time PCR machine (Applied Biosystem, Foster City, California, USA). For this analysis, we use Taq primer assay which had rs number 1143627 (Thermo Fisher Scientific, Waltham, California, USA). Reverse and forward primer sequences were used defining used for possible mutations in target variations
Visual Analog Scale - Pain Assessment | baseline
  Visual Analog Scale (VAS) was used to assess the pain severity of the patients. According to VAS, for pain intensity, it is generally rated as "no pain" 0 points and "moderate pain"5, worst pain imaginable" as 10 points (100 mm scale). They were asked to mark their average pain levels by considering one week. The pain level was questioned separately during resting and activity.
Oswestry Disability Index - Functional Disability | baseline
  The functional level assessment was evaluated using the Oswestry Disability Index (ODI). This scale is preferred to measure the performance of the activities necessary for daily living and to define their limitations. In this scale, consist of 10 sections are included about pain level, inactivity daily living, heavy lifting, walking, sitting, standing, sleeping, sexual life, social life and travelling. There are 6 options in each question, and the patient is asked to choose the expression of his condition.
The Range of Motion of the lumbar spine | baseline
  Physiotherapist will measure the Range of Motion of the lumbar spine by using digital goniometer
Modified Schober Test - Lumbar Spine Flexibility | baseline
  Physiotherapist will measure. The posterior interval between both spina iliaca was marked for measurement. After determining 10 cm above and 5 cm below the marked area, the patient was asked to perform trunk flexion while standing. The difference between the initial value and is noted in cm. The difference of 0-5 cm in the test shows that the flexion flexibility decreases, and the difference over 10 cm shows that the flexibility increases. Values between 5-10 cm are considered normal.

SECONDARY OUTCOMES:
Pfirrmann's grading - Total Disc Degenerative Disc Score | baseline
  Lumbar sagittal Magnetic Resonance Imaging (MRI) was used for the analysis of disc degeneration, and herniation and sections of 5 mm thick were taken. T2-weighted MR examinations of all cases included in the study, independently by a radiologist who is blind to the clinical condition of the cases it was evaluated. Disc degeneration graded according to Pfirrmann's grading. For each case, all lumbar discs were scored individually (L1-2, L2-3, L3-4, L45, L5-S1) total score was calculated.
McNab's disc classification - Disc displacements | baseline
  Lumbar sagittal Magnetic Resonance Imaging (MRI) was used for the analysis of disc displacements.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ünsal, M.S.c, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No